CLINICAL TRIAL: NCT02149706
Title: A Phase IIb Study of NeuroVax™, a Novel Therapeutic TCR Peptide Vaccine for SPMS of Multiple Sclerosis Slowing Disease Progression Via Vaccination
Brief Title: A Study of NeuroVax™, a Novel Therapeutic TCR Peptide Vaccine for SPMS of Multiple Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Immune Response BioPharma, Inc. (Industry)
Collaborators: cro (Ambiguous)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Immune Response 2020
Record Dates: First submitted 2014-05-24; First posted 2014-05-29 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Multiple Sclerosis
Keywords: Secondary Progress Multiple Sclerosis; SPMS; Multiple Sclerosis; NeuroVax
MeSH Terms: conditions — Multiple Sclerosis | interventions — NeuroVax vaccine; HIV-1 immunogen, incomplete Freund's adjuvant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NeuroVax (Experimental): NeuroVax
  Interventions: Biological: NeuroVax
- IFA Incomplete Freund's Adjuvant (Placebo Comparator): Incomplete Freund's Adjuvant IFA
  Interventions: Biological: IFA Incomplete Freund's Adjuvant

INTERVENTIONS:
Biological: NeuroVax — NeuroVax consists of a Trivalent TCR Peptide Formulation in IFA
  Arms: NeuroVax
Biological: IFA Incomplete Freund's Adjuvant — IFA Placebo Incomplete Freund's Adjuvant
  Arms: IFA Incomplete Freund's Adjuvant

SUMMARY:
Multi-center, randomized , double-blind, placebo-controlled , two arm parallel design study of NeuroVax™ vs. Incomplete Freund's Adjuvant ( I F A) placebo. 150 subjects with Secondary Progressive SPMS.

DETAILED DESCRIPTION:
The primary objective is to compare between treatment groups the Measures of neurologic disability EDSS scores.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 18 Years to 70 Years
* Genders Eligible for Study: Both
* Accepts Healthy Volunteers: No Criteria
* Subject is between 18 and 70 years of age, inclusive.
* Definite MS by the revised McDonald criteria (2005) (Appendix A), with a Secondary Progressive course.
* Expanded Disability Status Scale (EDSS) >=score 3.5 (Appendix B).
* Two or more documented clinical relapses of MS in the preceding 24 months OR one documented clinical relapse of MS in the preceding 1 2 months prior to screening .
* Laboratory values within the following limits:
* Creatinine 1 . 5 x high normal.
* Hemoglobin

Exclusion Criteria:

* Subjects currently prescribed Campath or Lemtrada

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-03-09 (Estimated); Primary Completion 2022-03-09 (Estimated); Study Completion 2022-03-09 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to compare between treatment groups the Measures of neurologic disability EDSS score | 48 Weeks
  The primary objective is to compare between treatment groups the Measures of neurologic disability EDSS scores improvements

SECONDARY OUTCOMES:
Secondary measurements objectives immunologic evaluations | 48 Weeks
  Secondary measurements objectives immunologic evaluations increases in white blood cell counts & FOXP+3 expression increases

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Bartholomew, Ph.D, Study Director — Immune Response BioPharma, Inc.
Locations (1):
- CRO, San Diego, California, United States